CLINICAL TRIAL: NCT04619875
Title: A Randomized, Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect of Increasing Intake Amounts of Two Novel Glycans on the Gut Microbiota of Healthy Subjects
Brief Title: A Clinical Study to Assess the Effect of Increasing Intake Amounts of Two Novel Glycans on the Gut Microbiota of Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K008-117
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Microbiome; Kaleido; Kaleido Biosciences; Oligosaccharide; Glycan; Microbiome Metabolic Therapy; KB174; KB5; SG1
MeSH Terms: interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactulose (Other)
  Interventions: Other: Lactulose
- KB5 (Other)
  Interventions: Other: KB5
- SG1 (Other)
  Interventions: Other: SG1

INTERVENTIONS:
Other: KB5 — KB5, a novel glycan, is a Kaleido laboratory code for KB174
  Arms: KB5
Other: SG1 — SG1 is a novel glycan
  Arms: SG1
Other: Lactulose — Lactulose is a synthetic dissacharide
  Arms: Lactulose

SUMMARY:
This exploratory, randomized, open label study aims to explore the safety, tolerability, pharmacokinetics, and effects of increasing intake amounts of two novel glycans on the gut microbiota of healthy subjects.

ELIGIBILITY:
To be eligible for inclusion, the patient must fulfill all of the following criteria at screening:

* Able and willing to provide informed consent
* Willing to provide multiple stool samples
* Be male or female, ≥18 and ≤65 years of age
* Have a body mass index ≥20 and <40 kg/m2
* No current renal, hepatic or metabolic disease, significant dyslipidemia, or infection.
* Willing to adhere to dietary requirements as stated in the protocol.
* Willing to continue his/her normal diet and exercise routine.
* Willing to continue taking any current supplements and vitamins, (with the exception of prebiotic or probiotic supplements) that the subject is currently taking, for the duration of the study.
* Negative urine drug screen
* If subject is female, have a negative urine pregnancy test at Screening and be willing to engage in method of contraception until completion of the study

Patients will be excluded from the study if they meet any of the following criteria at screening:

* Currently taking probiotic or prebiotic dietary supplements, or have taken them in the past 28 days (prior to Screening Visit), or unwilling to avoid probiotic or probiotic dietary supplements for the duration of the study
* Currently taking, or have taken in the last 7 days, drugs or other compounds to modulate gastrointestinal motility
* Recent history (within six weeks of Screening) of the following conditions requiring medical attention or treatment, including over-the-counter medications: constipation, diarrhea, and/or acute GI illness.
* Systemic antibiotics taken within the previous three months (prior to Screening Visit).
* History of or active inflammatory bowel disease
* History of or active irritable bowel syndrome
* History of or active autoimmune disease
* History of or active GI malignancy
* Established pre-diabetic status (eg, multiple fasting blood glucose measurements 100 to 125 mg/dL inclusive, or history of failed glucose tolerance tests) and as assessed by HbA1c test
* Have used an investigational drug or device within 30 dyas of study or be concurrently enrolled in another investigational drug or device study within 30 days of the study (prior to the Screening Visit)
* Subject is a current smoker
* Subject has a history of drug and/or alcohol abuse
* Contraindications, sensitivity, or known allergy to the use of the study product(s) or their components
* Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study (prior to the Screening Visit)
* Individuals who, in the opinion of the PI, are considered to be poor attendees or unlikely for any reason to be able to comply with the study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by incidence of adverse advents | Day -8 to Day 35
Tolerability as assessed by Gastrointestinal Tolerability Questionnaire (GITQ) score | Day -8 to Day 35
  The GITQ is an assessment of the frequency and severity of GI symptoms, eg., gas, abdominal pain, calculated on a scale from 0 (None/Not applicable) to a maximum score of 60 (Severe/Much more than usual) for all questions
Tolerability as assessed by change in Bristol Stool Scale (BSS) | Day -8 to Day 35
  The BSS is an assessment of stool consistency on a scale from 1 (separate hard lumps, like nuts, hard to pass) through 7 (watery, no solid pieces, entirely liquid)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (1):
- Biofortis, Addison, Illinois, United States